CLINICAL TRIAL: NCT04680663
Title: Peripheral Perfusion Index Versus Serum Lactate Levels as Predictor of Postoperative Complications and Prolonged ICU Stay After Lengthy Surgical Procedures: a Prospective Observational Study
Brief Title: Predictor of Postoperative Complications After Lengthy Noncardiac Surgery
Acronym: complication
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Assistant Professor of Anesthesia, Pain management and Surgical ICU, Cairo University
Other Study IDs: MS-390-2020
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non complications group: where the non-complicated patients is the patients running the normal postoperative course of surgery and without any need for intervention
  Interventions: Diagnostic Test: Peripheral Perfusion index; Diagnostic Test: serum lactate level
- complications group: any deviation from the normal post-operative course
  Interventions: Diagnostic Test: Peripheral Perfusion index; Diagnostic Test: serum lactate level

INTERVENTIONS:
Diagnostic Test: Peripheral Perfusion index — Peripheral Perfusion index is the ratio between pulsatile blood flow to non pulsatile blood flow or static blood in the peripheral tissue
Diagnostic Test: serum lactate level — Blood lactate (product of metabolism) level is maintained by a cycle of continuous production and metabolism allowing it to be kept within normal values

SUMMARY:
Many patients undergoing long time surgery will manifest increased level of blood lactate.

Hyperlactacidemia can cause disturbance of internal environment, then leading to increased complications and longer ICU stay, even death. For postoperative patients, we must ensure adequate perfusion in order to minimize the length of hyperglycemia and improve patients' outcomes. With regard to lactate, it provides information about prefusion, but not timely enough for its delay on reflecting hypoperfusion. And it's not real-time and non-invasive.

Peripheral perfusion index (PPI) is an indicator reflecting hypoperfusion in critical patients. It is measured using pulse co-oximetry technology which is characterized by being real-time and noninvasive. PPI is defined as "the ratio of pulsatile blood flow to the non-pulsatile blood flow", mirroring the strength of blood flow and quality of perfusion at sensor site, reflecting perfusion state of the body part . In contrast to lactate value, it's real-time and easy to monitor.

ELIGIBILITY:
* Inclusion criteria
* Adult patients above 18 years of age.
* Both genders
* surgical time planned to be > 120 minutes .
* surgical time predicted to exceed the planned time and prolongation of surgical time > 120 minutes occured will be included in the study .
* ASA physical status of I-II
* Patients scheduled for elective surgery under general anaesthesia .
* Exclusion criteria
* Refused to participate .
* patient with disease affecting blood flow to the hands where probe will be applied .
* patient with hand injuries so probe cannot be applied
* Patient with sever renal and liver disease
* Discharging against medical advice or reported death during ICU stay at first 48 hours after ICU admission .
* Pregnancy or emergency surgery .
* shortening of the planned surgical time to be less than 120 minutes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be designed to recruit patients scheduled for elective surgery with duration > 120 minutes under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Peripheral perfusion index | up to 48 hours
  at end of surgery as early predictor of postoperative complications .
serum lactate level | up do 48 hours
  at end of surgery as early predictor of postoperative complications .

SECONDARY OUTCOMES:
serum lactate level | UP TO 30 day
  at end of surgery as early predictor of postoperative complications .
Peripheral perfusion index | UP TO 30 DAY
  at end of surgery as predictor seversity of postoperative complications .
Postoperative complications | up to 30 day
  the Clavien-Dindo classification system Grade I complications Grade II complications Grade III complications Grade IV complications
hemodynamic change | up do 48 hours
  mean arterial blood pressure
heart rate | up do 48 hours
  hemodynamic change

CONTACTS AND LOCATIONS:
Overall Officials: Amr s wahdan, MD, Principal Investigator — Cairo university , Cairo, Egypt
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided